CLINICAL TRIAL: NCT05690802
Title: Palonosetron Hydrochloride Capsules (Ruoshan ®) Used to Prevent and Control Chemotherapy for Tumor Patients Real World Study on the Safety of Nausea and Vomiting Reduction
Brief Title: The Safety and Effectiveness of Palonosetron Hydrochloride Capsule Was Used to CINV
Acronym: TSEPHCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQXB-R-001
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Palonosetron

STUDY DESIGN:
Intervention Model Description: Palonosetron hydrochloride capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palonosetron hydrochloride capsules (Experimental): The recommended dose for adults is 0.5mg (1 capsule) for a single oral dose about 1 hour before chemotherapy.
  Interventions: Drug: Palonosetron hydrochloride capsules

INTERVENTIONS:
Drug: Palonosetron hydrochloride capsules — This protocol only stipulates "Palonosetron capsule containing hydrochloric acid protocol", and does not make uniform provisions on the treatment course, and does not interfere with the actual clinical usage and dosage.
  Other Names: Ruoshan ®

SUMMARY:
To observe and evaluate the safety and effectiveness of Palonosetron hydrochloride capsule in preventing acute nausea and vomiting caused by moderate emetic chemotherapy; The characteristics of the applicable population, clinical medication and clinical benefits of Palonosetron Hydrochloride Capsules were analyzed.

DETAILED DESCRIPTION:
At present, as the mainstream antiemetics of CINV, oral administration is the most commonly used method of drug therapy. Clinical studies showed that there was no difference in the efficacy of 5-HT3 receptor antagonist between different administration routes (oral and intravenous). At the same time, because the oral route is the most convenient, oral preparations provide more and more convenient choices for clinicians and patients. To observe and evaluate the safety and effectiveness of Palonosetron hydrochloride capsule in preventing acute nausea and vomiting caused by moderate emetic chemotherapy; The characteristics of the applicable population, clinical medication and clinical benefits of Palonosetron Hydrochloride Capsules were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* For patients with malignant tumors who can accept chemotherapy, the disease type is not limited. The specific chemotherapy scheme is the chemotherapy scheme with moderate risk of vomiting (for the risk level of vomiting, refer to the 2019 CSCO anti-tumor treatment related nausea and vomiting prevention and treatment guidelines);
* 18-75 years old, KPS score ≥ 70, and the expected survival time is more than 3 months;
* Before treatment, ECG, blood routine test, liver and kidney functions and electrolytes were basically normal;
* All patients signed the informed consent form

Exclusion Criteria:

* Patients with chemotherapy contraindications, patients allergic to 5-HT3RA, pregnant women and lactating women;
* People with digestive tract obstruction; Patients with serious heart disease, liver and kidney disease and metabolic disorder; Patients suffering from epilepsy or using psychotropic and sedative drugs;
* Used antiemetic drugs or chemicals within 24 hours.Those who have vomited before treatment may have brain metastasis, intracranial hypertension, gastrointestinal obstruction, psychological abnormalities, etc.Patients with factors causing nausea and vomiting.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Any adverse event after treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hong, master, Study Chair — Air Force Military Medical University, China
Locations (1):
- The First Affiliated Hospital, the Air Force Medical University, Xi'an, Shaan'xi, China